CLINICAL TRIAL: NCT01112540
Title: Morphine in Acute Abdominal Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Akdeniz University (Other)
Other Study IDs: RCT_AE_02
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Abdominal Pain
Keywords: to evaluate the anal. efficacy of IV morph. vs. place. for elderly presenting to the ED with UAP and determine if it has an impact on diag. accu. and phy. exam
MeSH Terms: conditions — Abdominal Pain | interventions — Morphine

ARMS (2):
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Morphine
- Morphine (Experimental)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — 0.1 mg/kg Intravenous bolus

SUMMARY:
The investigators primary outcome measure was the clinically important change in diagnostic accuracy and physical examination in the morphine vs. placebo group. After follow up information was obtained and patients data were recorded on the SPSS data chart, two blinded coauthors (general surgeon and emergency physician) determined the clinically important diagnostic accuracy and change in physical examination. They firstly defined clinically important diagnostic errors, as any disagreement between the preliminary and final diagnosis that might be expected to have adverse effect on the patient's general status. If coauthors decided an instance of diagnostic error as clinically important, this was coded "diagnostic discordance" for statistical analysis. While the preliminary diagnosis was determined as accurate or not different from the final diagnosis, this was coded "diagnostic accuracy" for statistical analysis. Secondary outcome measures included the need for rescue drugs at 30 minutes, the presence of at least one adverse event, demographic features and final diagnosis of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Elderly (65 years or older) patients with non-traumatic UAP of less than 48 hours' duration were included in the study. Participants were required to have a UAP and report either "mild" or greater pain intensity on a four-point verbal rating scale (VRS) or at least 20 mm on a 100 mm visual analogue scale (VAS).

Exclusion Criteria:

* Exclusion criteria included known allergy or contraindication to morphine, or any opioid analgesic
* Hemodynamic instability (systolic blood pressure less than 100 mm-Hg)
* Use of any analgesic within 6 hours before ED presentation
* Patients refused to participate to the study
* Incooperated to the VAS
* Isolated flank pain or previous study enrollment
* Patients with known renal, pulmonary, cardiac or hepatic failure were also excluded.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult

PRIMARY OUTCOMES:
Our primary outcome measure was the clinically important change in diagnostic accuracy and physical examination in the morphine vs. placebo group.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)